CLINICAL TRIAL: NCT01350583
Title: A Pilot Study of Oral Bicarbonate as Adjuvant for Pain Reduction in Patients With Tumor Related Pain
Brief Title: Bicarbonate for Tumor Related Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Left Moffitt
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-16047
Record Dates: First submitted 2011-05-06; First posted 2011-05-10 (Estimated); Results first posted 2013-08-08 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-06

CONDITIONS: Neoplasm Related Pain (Acute) (Chronic)
Keywords: tumor related pain
MeSH Terms: conditions — Cancer Pain | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sodium Bicarbonate Therapy (Experimental): Dose Escalation
  Interventions: Drug: Sodium Bicarbonate (NaHCO3)

INTERVENTIONS:
Drug: Sodium Bicarbonate (NaHCO3) — Treatment consisted of 0.15 g/kg/day Sodium Bicarbonate (NaHCO3) increasing to 0.3 g/kg/day after 1 week if well tolerated. Further dose increment to 0.6 g/kg/day was to be done after 2 weeks of starting sodium bicarbonate if prior dose levels were well tolerated.

SUMMARY:
The purpose of this study is to:

* Determine how well people tolerated sodium bicarbonate taken by mouth in higher doses than those usually given for heartburn.
* Determine if sodium bicarbonate can reduce cancer-related pain. Right now, the investigators do not know for sure if these higher doses will be well tolerated or if they will reduce the pain associated with cancer. The investigators are doing this study to see if sodium bicarbonate is well tolerated and if it can reduce the requirements for pain medications.

DETAILED DESCRIPTION:
The study is a single institution, non-randomized, single arm pilot study to evaluate the efficacy of adjuvant therapy with sodium bicarbonate for tumor related pain. Patients will receive sodium bicarbonate (0.15 g/kg/day for 1 weeks and if tolerated 0.3 g/kg/day for one week and if this dose is tolerated 0.6 g/kg/day) for 4 weeks. The sodium bicarbonate will be provided to the patient as a powder and consumed after it is mixed with about 250 cc (about 1 cup) of water. In consultation with the PI, the patients will be permitted to mix the sodium bicarbonate with a commercially available drink instead of water provided the liquid has an acid/base balance (pH) of 7.4 or greater. Patients with a good tolerance to study therapy and with at least a 30% improvement in pain intensity (by VAS) compared to baseline after 3 weeks of therapy and who wish to continue study therapy will be allowed to continue sodium bicarbonate therapy under the direction of their treating physician. Patients without at least a 30% improvement in pain intensity at 3 weeks will discontinue study therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic or unresectable solid malignancy or hematologic malignancy (multiple myeloma or lymphoma) and must have moderate to severe tumor related pain (VAS>4) on a stable opioid regimen (at least 3 days of an opiate regimen).
* No planned palliative surgery, palliative radiotherapy for at least 2 weeks. However prior radiotherapy, and surgery is allowed and not limited to the number of procedures and courses. Concomitant chemotherapy is allowed. In addition, when it is anticipated that chemotherapy may result in rapid pain relief (less than 2 weeks), patients will only be enrolled after completing their first cycle of chemotherapy and provided their pain level is greater than 4 on the VAS.
* No evidence of neurologic or psychiatric compromise which in the opinion of the investigator will interfere with completion of study assessments
* Life expectancy greater than 3 months
* Age greater than 18 years and able to understand and sign the informed consent document
* Patients must have an Eastern cooperative oncology group (ECOG) performance status less than 4.

Exclusion Criteria:

* Patients with neuropathy and/or neuropathic pain as the only pain syndrome are not eligible. Patients with chronic non malignant pain are not eligible.
* Patients with renal insufficiency (creatinine > 2.5 mg/dL) are excluded
* Patients with history of congestive heart failure or pulmonary artery hypertension will be excluded
* Any patient who in the opinion of the investigator is dehydrated at the time of initial evaluation will be excluded.
* Patients with uncontrolled hypertension (systolic pressure >140, diastolic pressure >90) despite maximal antihypertensive therapy.
* Patients unable to ingest of oral sodium bicarbonate (such as patients with dysphagia or severe nausea)
* Patients with ECOG performance status 4
* Patients with acute leukemia, myelodysplastic syndrome, and chronic myeloid leukemia are not eligible.
* Pregnant or lactating patients are not eligible.
* Patients with estimated survival less than 3 months
* Patients with known allergy to sodium bicarbonate or patients with preexisting renal or acid base disorders for which sodium bicarbonate is contraindicated (such as metabolic alkalosis, severe congestive heart failure, hypernatremia, and hypocalcemia [see above]).
* Patients with severe ongoing infections which places the patients at increased risks from therapy in the opinion of the investigator.
* Patients who are receiving and or will receive, during their participation in study, an oral chemotherapeutic agent whose bioavailability could be altered by the ingestion of sodium bicarbonate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gillies, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Gillies RJ, Ibrahim-Hashim A, Ordway B, Gatenby RA. Back to basic: Trials and tribulations of alkalizing agents in cancer. Front Oncol. 2022 Nov 14;12:981718. doi: 10.3389/fonc.2022.981718. eCollection 2022. PMID 36452492

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to enrollment at Moffitt Cancer Center from August, 2010 through July, 2011. Two participants were actually enrolled during 2010.
Groups:
- Sodium Bicarbonate Therapy: Dose Escalation
  Sodium Bicarbonate (NaHCO3) : Treatment consisted of 0.15 g/kg/day Sodium Bicarbonate (NaHCO3) increasing to 0.3 g/kg/day after 1 week if well tolerated. Further dose increment to 0.6 g/kg/day was to be done after 2 weeks of starting sodium bicarbonate if prior dose levels were well tolerated.
Period: Overall Study
Arm/Group | Sodium Bicarbonate Therapy
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sodium Bicarbonate Therapy
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With Improvement
Description: Percent of patients with greater than 30% improvement in pain intensity by visual assessment scale.
Time Frame: 4 weeks per participant
Population: Results data was not calculated due to low accrual. Outcome Measures were based on 25 evaluable participants. That goal was not reached.
Arm/Group | Sodium Bicarbonate Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Percent of Patients Where Treatment Was Well Tolerated
Description: Tolerability and safety of oral sodium bicarbonate in patients with moderate to severe tumor related pain
Time Frame: 4 weeks per participant
Population: Results data was not tabulated due to low accrual. Outcome Measures were based on 25 evaluable participants. That goal was not reached.
Arm/Group | Sodium Bicarbonate Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Improvement in Pain Indices
Description: Improvement in pain indices (Memorial Symptom Assessment Scale, MSAS) and Brief Pain Inventory (BPI).
Time Frame: 4 weeks per participant
Population: as for outcome 2
Arm/Group | Sodium Bicarbonate Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Sodium Bicarbonate Therapy
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Bicarbonate Therapy (N=2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema: head and neck (Blood and lymphatic system disorders) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 1 (3)
Pain - Head/headache (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This Pilot Supportive Care study ended prematurely due to slow accrual and the initiating principal investigator leaving the institution. The outcome measures were based on 25 evaluable participants and there were only 2 participants enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes